CLINICAL TRIAL: NCT03872193
Title: Effects of Virtual Reality on Transtibial Amputation Ouality of Life,Performance, Balance,Prothesis Adaptation and Gait Outcomes
Brief Title: Effects of Virtual Reality on Transtibial Amputation Physiotherapy Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatih Erbahceci, Clinical Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Virtual Reality Physiotherapy
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Virtual Reality
Keywords: Amputation; Virtual Reality; Rehabilitation
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: One group only physiotherapy second group takes physiotherapy and virtual reality exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physio Therapy (Experimental): We intervention this group some routine exercises. They had balance exercises, gait training,incline surface gait,bloked surface gait training and recreational activities. Extremity strengthenin exercises,balance exercises and increasing endurance are applied for this amputees.
  Interventions: Other: Exercise
- Virtual Reality (Experimental): This group had physical therapy program plus virtual reality exercises. They had balance exercises, gait training,incline surface gait,bloked surface gait training and recreational activities. Extremity strengthenin exercises,balance exercises and increasing endurance are applied for this amputees. And virtual reality exercises were done for this group. Skiing,kayak, football,rafting and jumping activities were done in this exerciese.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Virtual Reality Exercies

SUMMARY:
The aim of this study is to compare the effects of virtual reality applications on quality of life, performance, balance, prosthesis adaptation and gait parameters in individuals with transtibial amputation. 20 Transtibial amputee were included in study. All participants were using transtibial prothesis with active vacuum system at least 1 year. Participants were divided into two groups. While a group of virtual reality applications were being performed additionally standart physiotherapy, only standard physiotherapy methods were applied in the second group. Balance and gait practices were performed for each group. Individuals were treated for 3 days a week for 4 weeks, and individuals were evaluated before and after treatment. Individuals were evaluated for quality of life, performance, balance, prosthesis adaptation and time-distance parameters of walking.

DETAILED DESCRIPTION:
The aim of this study is to compare the effects of virtual reality applications on quality of life, performance, balance, prosthesis adaptation and gait parameters in individuals with transtibial amputation.20 transtibial amputee with 36 mean age were included in study. All participants were using transtibial prothesis with active vacuum system at least 1 year. Participants were divided into two groups. While a group of virtual reality applications were being performed, standard physiotherapy methods were applied in the second group. Balance and gait practices were performed for each group. Individuals were treated for 3 days a week for 4 weeks, and individuals were evaluated before and after treatment. Individuals were evaluated for quality of life, performance, balance, prosthesis adaptation and time-distance parameters of walking.

For this purpose, SF-36 Questionnaire, 6-minute walking test, one leg rest time, Trinity Amputation and Prosthetic Experience Scale, wearable biometric device and footprint method were utilized. There was a statistically significant difference between the two groups in pre-treatment and post-treatment performance, balance and gait parameters in the groups of individuals (p <0.05). The quality of life pain parameter was statistically decline in the group receiving virtual reality (p<0.05). On the other hand, significant differences in the quality of life and prosthesis adaptation of the individuals were not found between the groups (p> 0.05). The results of this study showed that virtual reality practices and standard physiotherapy methods are effective on performance, balance and walking in transtibial amputee rehabilitation. It is thought that it will be important to perform virtual reality applications in amputee rehabilitation separately in both methods, in addition to standard physiotherapy methods, to include in rehabilitation process, to bring an ability of alternative application to professionals working in this area and to work about amputees with using different suspension systems and with different amputation levels.

ELIGIBILITY:
Inclusion Criteria:

* transtibial and unilateral amputation
* At least 1 year prothesis usage, 18- 65 year age,
* At least 15 min independent walking ability,
* Stabile stump volume,
* Standart stump lentgh,
* Enough kognition for evaluation and tests.

Exclusion Criteria:

* walking and other activities to prevent; shortness of muscle, limitation of joint motion and phantom pain in stump, presence of any discomfort or systemic health problem that may affect the gait outside the amputation
* presence of visual problems to prevent participation in virtual reality applications,
* use of walking aids

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-07-10 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-06-10 (Actual)

PRIMARY OUTCOMES:
Quality of Life measured of individuals: SF-36 Scale | 10 minute
  SF-36 Quality of Life Scale, higher values represent a better
Balance Test | 5 minute
  Single Leg Balance Test,higher values represent a better
Performance Test | 6 minute
  6 minute walk test,higher values represent a better
Prothesis Satisfaction: Trinity Amputation Prothesis Experience Scale | 5 minute
  Trinity Amputation Prothesis Experience Scale; 5 point likert scale,5-75 point, activity limitation,physicosocial adaptation,prothesis satisfaction
Gait Parameters | 6 minute
  Wearable Biometric Device

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yildirim Sahan T, Erbahceci F. Effects of Virtual Reality on Transtibial Amputation Rehabilitation Outcomes: A Randomized Study. Games Health J. 2023 Dec;12(6):459-467. doi: 10.1089/g4h.2023.0052. Epub 2023 Nov 7. PMID 37934289
- [Derived] B Aledi L, Flumignan CD, Trevisani VF, Miranda F Jr. Interventions for motor rehabilitation in people with transtibial amputation due to peripheral arterial disease or diabetes. Cochrane Database Syst Rev. 2023 Jun 5;6(6):CD013711. doi: 10.1002/14651858.CD013711.pub2. PMID 37276273